CLINICAL TRIAL: NCT02242006
Title: Antimicrobial Pharmacokinetics in Critically Ill Adults During Sustained Low Efficiency Dialysis (SLED)
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 20140429
Record Dates: First submitted 2014-09-09; First posted 2014-09-16 (Estimated); Last update posted 2021-04-29 (Actual); Status verified 2014-09

CONDITIONS: Critical Illness; Kidney Injury; Pharmacokinetics
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- piperacillin/tazobactam: Serial serum sampling of patients receiving piperacillin/tazobactam and SLED simultaneously
  Interventions: Other: serial serum sampling for quantification of drug concentration
- meropenem: Serial serum sampling of patients receiving meropenem and SLED simultaneously
  Interventions: Other: serial serum sampling for quantification of drug concentration
- vancomycin: Serial serum sampling of patients receiving vancomycin and SLED simultaneously
  Interventions: Other: serial serum sampling for quantification of drug concentration

INTERVENTIONS:
Other: serial serum sampling for quantification of drug concentration

SUMMARY:
Severe acute kidney injury (AKI) is a common complication of critical illness affecting almost half of all patients with septic shock. Extracorporeal renal replacement therapy is a cornerstone in the management of AKI in these patients. Options for renal replacement therapy include continuous renal replacement (CRRT) therapy, intermittent dialysis (IHD) or a hybrid form of the two called sustained low efficiency dialysis (SLED). Globally there is a push to switch from traditional CRRT to SLED. Although there are resource and financial comparative benefits to SLED there is almost no literature describing how to dose antimicrobials (or other drugs for that matter). It appears that drug clearance on SLED may be more efficient than CRRT but not as efficient as IHD making extrapolation from these bodies of literature inappropriate for SLED. The investigators are proposing to conduct the population pharmacokinetic studies for the three most commonly used antimicrobials in critically ill patients receiving SLED therapy (piperacillin-tazobactam, meropenem and vancomycin). Population pharmacokinetic modeling of these drugs will provide estimates and sources of variability around pharmacokinetic parameters that will subsequently be used for Monte Carlo simulation to determine the most appropriate dosing regimens to achieve therapeutic targets while minimizing the risk of toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill adults [age ≥ 18] admitted to one of two of the medical/surgical intensive care units (ICUs) of The Ottawa Hospital, who require SLED and are or will receive meropenem, piperacillin-tazobactam or vancomycin therapy at any dose.

Exclusion Criteria:

* Patients for whom participation via the informed consent process is denied.
* Critically ill patients with a hypermetabolic state due to >25% coverage of body surface area burn, cystic fibrosis, spinal cord injury, bariatric patients (defined as >150kg total body weight)
* Patient is pregnant as per a positive serum or urine βHCG qualitative assay
* Patient does not have a closed-system arterial or central venous catheter (to minimize blood wastage)
* Patients receiving concomitant drugs known to interact with the metabolism or clearance of the antimicrobial of interest according to Micromedex 2.0 (Truven Health Analytics Inc 2013)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critically ill adults admitted to an ICU
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
drug clearance | During the first run of SLED after study inclusion
  Serial serum samples will be obtained after drug administration and during SLED to determine drug clearance during SLED.
volume of distribution | During the first run of SLED after study inclusion
  Serial serum samples will be obtained after drug administration and during SLED to determine drug volume of distribition during SLED.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada